CLINICAL TRIAL: NCT03930758
Title: Parameters of Exercise to Prevent Type 2 Diabetic Osteoporosis in Postmenopausal Women
Brief Title: Preventing Diabetic Osteoporosis With Exercise
Acronym: DIABETICBONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Wisconsin, La Crosse (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dr. Katarina Borer, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: HUM32227/ HUM32700; R15DK082800 (NIH); M01RR024986 (Other Grant/Funding Number: Michigan Institute of Clinical and Health Research)
Record Dates: First submitted 2019-04-19; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Study consisted of 5 experimental trials (or arms), of which 4 were compared to a sedentary (or control) arm. The five trials were: Uphill exercise before the meals (UBM), Uphill exercise after the meals (UAM), Downhill exercise before the meals (DBM), and Downhill exercise after the meals (DAM), and the Sedentary (Sed) or control trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Uphill exercise before the meals (Experimental): 40 minutes of uphill treadmill exercise at +6o slope completed 1 hour before eating the meal
  Interventions: Combination Product: Behavior intervention of uphill exercise; Combination Product: Dietary intervention of exercise before the meal
- Uphill exercise after the meals (Experimental): 40 minutes of uphill treadmill exercise at +6o slope started 1 hour after eating the meal
  Interventions: Combination Product: Dietary intervention of uphill exercise; Combination Product: Dietary intervention of exercise after the meal
- Downhill exercise before the meals (Experimental): 40 minutes of downhill treadmill exercise at -6o slope completed 1 hour before eating the meal
  Interventions: Combination Product: Behavior intervention of downhill exercise; Combination Product: Dietary intervention of exercise before the meal
- Downhill exercise after the meals (Experimental): 40 minutes of downhill treadmill exercise at -6o slope started 1 hour after eating the meal
  Interventions: Combination Product: Behavioral intervention of downhill exercise; Combination Product: Dietary intervention of exercise after the meal
- Sedentary trial (Sham Comparator): A trial with no exercise
  Interventions: Combination Product: Behavioral intervention of sedentary no-exercise trial; Combination Product: Dietary intervention of eating two meals

INTERVENTIONS:
Combination Product: Behavior intervention of uphill exercise — 40 minutes of uphill exercise
  Arms: Uphill exercise before the meals
Combination Product: Dietary intervention of exercise before the meal — 40 minutes of uphill exercise completed 1 h before the meal
  Arms: Uphill exercise before the meals
Combination Product: Dietary intervention of uphill exercise — 40 minutes of uphill exercise
  Arms: Uphill exercise after the meals
Combination Product: Dietary intervention of exercise after the meal — 40 minutes of uphill exercise started 1 hour after gthe meal
  Arms: Uphill exercise after the meals
Combination Product: Behavior intervention of downhill exercise — 40 minutes of downhill exercise
  Arms: Downhill exercise before the meals
Combination Product: Dietary intervention of exercise before the meal — 40 minutes of downhill exercise completed 1 hour before the meal
  Arms: Downhill exercise before the meals
Combination Product: Behavioral intervention of downhill exercise — 40 minutes of downhill exercise
  Arms: Downhill exercise after the meals
Combination Product: Dietary intervention of exercise after the meal — 40 minutes of downhill exercise started 1 hour after the meal
  Arms: Downhill exercise after the meals
Combination Product: Behavioral intervention of sedentary no-exercise trial — Sedentary no-exercise trial
  Arms: Sedentary trial
Combination Product: Dietary intervention of eating two meals — Meals eaten at 10 and 17 h during a sedentary trial
  Arms: Sedentary trial

SUMMARY:
The two specific aims of the study were to determine whether:

1. Greater mechanical loading of downhill exercise will increase the osteogenic index (ratio between CICP, the marker of bone formation (c-terminal propeptide of type I collagen, and CTX, the marker of bone resorption (c terminal telopeptide of type I collagen)) to a greater extent than uphill exercise that provides lower ground-reaction force;
2. Exercise after the meals will induce greater osteogenic response than exercise pefore the meals as it is known that meal eating during daytime inhibits bvone resorption markers.

DETAILED DESCRIPTION:
The study addresses the problem that postmenopausal women with type 2 diabetes have a higher incidence of bone breaks despite their often normal bone mineral density (BMD).

The investigators pursued two hypotheses, that:

1. 40-minute bout of downhill exercise will increase the CICP/CTX osteogenic index to a greater extent than the same amount of uphill exercise; and
2. Performing exercise one hour after the meals will be more osteogenic than exercise before the meals.

Subjects were 15 postmenopausal women with type 2 diabetes, age 57.7 years, BMI 27.2 kg/m2 who were randomly assigned to two out of 5 trials:

Uphill exercise before the meals (UBM), Uphill exercise after the meals (UAM), Downhill exercise before the meals (DBM), Downhill exercise after the meals (DAM), and Sedentary, no-exercise, trial (SED). All subjects signed an informed consent approved by the University of Michigan Medical School Institutional Review Board. Subjects had their BMD measured with DXA at the outset.

Weight-maintenance meals contained 50% carbohydrate, 15% protein, and 25% fat and were provided at 10 h and 17 h. Exercise (40 minutes at 50% of maximal effort) on either uphill (+6o slope) or downhill treadmill (-6o slope) was performed either before the two meals, at 9 h and 16 h, respectively, or after the meals. at 11 h and 18 h, respectively.

Blood was drawn through an intravenous catheter from ante-cubital vein at hourly intervals between 8 and 20 h with two additional blood draws at 0 h and 6 h the next morning. Blood was treated with protease inhibitors, and plasma, frozen at -80o C, was used to measure bone markers, CICP, CTX, osteocalcin , and bone-specific alkaline phosphatase using Millipore chemoluminescen reagents, glucose by glucose oxidase, and hormones insulin, cortisol, parathyroid hormone (PTH) , and growth hormone (GH) by radio-immunoassays..

Mixed-model ANOVA was used for analysis of outcome measures where the trial procedures served as fixed variable and individual subjects as intercept variables.

ELIGIBILITY:
Inclusion Criteria:

postmenopausal type-2 diabetes melllitus age between 50 and 65 exercise less than 20 minutes three times a week

Exclusion Criteria:

metabolic disease other than type-2 diabetes and hormonally-corrected hypothyroidism musculo-skeletal disability that would preclude exercise smoker do not meet inclusion criteria

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10-08 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-20 (Actual)

PRIMARY OUTCOMES:
C-terminal propeptide of type I collagen | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of c-terminal propeptde of type 1 collagen (ng/ml)
C-terminal telopeptide of type 1 collagen | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of c-terminal telopeptide of type 1 collagen (ng/ml)
Osteocalcin | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of osteocalcin (ng/ml)
Bone-specific alkaline phosphatase | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of bone-specific alkaline phosphatase (ng/ml)

SECONDARY OUTCOMES:
Insulin | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of insulin (µU/ml)
Parathyroid hormone | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of parathyroid hormone (ng/ml)
Cortisol | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of cortisol (m/L)
Growth hormone | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of growth hormone (ng/ml)
Glucose | Hourly over 12 hours from the start of the trial, then at 16 hours, and at 22 hours, after the start of the trial
  Change over time in plasma concentration of glucose (mg/dl)
Dual-energy X-ray radiography | A week prior to the study baseline
  Whole-body dual-energy X-ray radiography scan
Novel Pedar | During two one-hour bouts of the exercise intervention
  Mechanosensitive shoe inserts for measurement of ground reaction force

CONTACTS AND LOCATIONS:
Overall Officials: Katarina T Borer, Principal Investigator — Professor Emerita